CLINICAL TRIAL: NCT03073395
Title: Preliminary Investigation of Uptake in PSMA Expressing Cancer, Biodistribution and Excretion of the Novel Radio Tracer [68Ga]P16-093 by PET/CT
Brief Title: Preliminary Evaluation of Uptake of [68Ga]P16-093 in Metastatic Prostate and Renal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 511-0003-A
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Renal Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dynamic group (Experimental): Dynamic imaging of suspected metastatic lesions with the investigation drug [68Ga]P16-093 in patients with a history of histologically confirmed cancer.
  Interventions: Drug: [68Ga]P16-093
- Biodistribution group (Experimental): Whole body imaging to determine human dosimetry of the investigational drug [68Ga]P16-093
  Interventions: Drug: [68Ga]P16-093

INTERVENTIONS:
Drug: [68Ga]P16-093 — Imaging by Positron Emission Tomography after iv injection of [68Ga]P16-093

SUMMARY:
An phase I study to evaluate the uptake of [68Ga]P16-093 in known or suspected metastatic prostate or renal cancer to establish the feasibility of using [68Ga]P16-093 to image PSMA expressing cancer. Measurement of the whole body biodistribution of [68Ga]P16-093 in prostate cancer patients post primary curative-intent treatment with stable PSA to generate human radiation dosimetry data.

ELIGIBILITY:
DYNAMIC GROUP:

Inclusion Criteria:

1. Participants will be male ≥ 18 years of age
2. History of histologically confirmed cancer that meets criteria for either a) or b)

   1. Prostate cancer with known or suspected recurrent or metastatic disease based on clinical imaging (e.g. CT, bone scan, MRI, ultrasound, FDG PET/CT, FACBC PET/CT) within 12 months of screening. If subject is post curative-intent local treatment (e.g. radical prostatectomy, local radiotherapy, brachytherapy) they must have had no intervening change in cancer treatment.

      OR
   2. Renal Cell cancer with known or suspected metastatic disease based on clinical imaging (e.g. CT, bone scan, MRI, ultrasound, FDG PET/CT)
3. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Estimated creatinine clearance (eGFR) < 30 mL/min (calculated from serum creatinine result within 30 days of screening)
2. Chemotherapy or radiation therapy within 2 weeks of screening
3. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
4. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful completion of the study

BIODISTRIBUTION GROUP:

Inclusion Criteria:

1. Participants will be male ≥ 18 years of age
2. History of prostate cancer that is post curative-intent local treatment (e.g. radical prostatectomy, local radiotherapy, brachytherapy) with clinical PSA levels that meet one of the following criteria

   1. Post-Prostatectomy (with or without adjuvant RT): PSA level that is < 0.2 ng/mL measured over at least 2 consecutive tests OR
   2. Post-Radiotherapy: PSA level that has not risen from nadir measured over at least 2 consecutive tests
3. If clinical imaging (e.g. bone scan, CT, MRI, ultrasound, PET/CT) has been done within 3 months of screening as part of standard clinical surveillance it must be negative or equivocal for sites of recurrent or metastatic disease (clinical imaging is not required for enrollment)
4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

1. Estimated creatinine clearance (eGFR) < 30 mL/min (calculated from serum creatinine result within 30 days of screening)
2. Androgen deprivation therapy (ADT) within 3 months prior to screening
3. Chemotherapy or radiation therapy within 2 weeks of screening
4. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
5. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful completion of the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Uptake of [68Ga]P16-093 in metastatic prostate and renal cancer | 0.5 - 3 hours after injection
  Standard uptake value (SUV) of [68Ga]P16-093 in apparent lesions detected by PET/CT.
Radiation dosimetry of [68Ga]P16-093 in patients with a history of prostate cancer | up to 3 hours after injection
  Radiation dosimetry (organ absorbed dose and effective dose) will be determined using region of interest data drawn on sequential PET/CT images and data from blood and / or urine obtained during scanning.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No